CLINICAL TRIAL: NCT06504719
Title: Safety and Efficacy Real-world Data of Trastuzumab Deruxtecan and Sacituzumab Govitecan in Patients With Advanced Breast Cancer
Brief Title: Safety and Efficacy Real-world Data of Trastuzumab Deruxtecan and Sacituzumab Govitecan
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE 11 ADC/23
Record Dates: First submitted 2024-04-09; First posted 2024-07-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: Trastuzumab deruxtecan; Sacituzumab govitecan; Efficacy; Safety; Brain metastasis; ILD
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Brain Neoplasms | interventions — Immunoconjugates; trastuzumab deruxtecan; sacituzumab govitecan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with trastuzumab deruxtecan or sacituzumab govitecan: Patients with TNBC, HER2-positive and/or hormone receptor positive advanced breast treated with trastuzumab deruxtecan or sacituzumab govitecan
  Interventions: Drug: Antibody-Drug Conjugates

INTERVENTIONS:
Drug: Antibody-Drug Conjugates — Patients with advanced breast cancer treated with ADCs
  Other Names: trastuzumab deruxtecan; Sacituzumab govitecan

SUMMARY:
The study aims to evaluate real-world efficacy and toxicity data of treatment with Trastuzumab deruxtecan (T-DXd), a HER2-targeting ADC and sacituzumab govitecan (SG), a TROP-2-targeting ADC in pretreated patients with advanced breast cancer.

DETAILED DESCRIPTION:
Antibody-drug conjugates (ADCs) have significantly changed the therapeutic landscape of advanced breast cancer. Trastuzumab deruxtecan (T-DXd), a HER2-targeting ADC and sacituzumab govitecan (SG), a TROP-2-targeting ADC, recently demonstrated superior efficacy over standard of care treatments depending on breast cancer subtype. The study aims to evaluate real-world efficacy and toxicity data of treatment with T-DXd and SG in pretreated patients with advanced breast cancer.

This study includes a retrospective/prospective multicenter review of medical records of patients with advanced breast cancer who received treatment with T-DXd and SG at Departments of Oncology, affiliated with the Hellenic Cooperative Oncology Group (HeCOG).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic/recurrent breast cancer
* 18 years of age
* Triple-negative (TNBC), HER2-positive and/or hormone receptor positive advanced breast cancer
* Treatment with an ADC at any of line of treatment
* Treatment with at least one cycle of T-DXd and/or SG

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients with histologically confirmed metastatic/recurrent breast cancer. Patients need to have received treatment with T-DXd and/or SG at Departments of Oncology in Departments of Oncology associated with the Hellenic Cooperative Oncology Group (HeCOG). Eligible patients are 18 years or older, diagnosed with triple-negative (TNBC), HER2-positive and/or hormone receptor positive advanced breast cancer, who received an ADC at any of line of treatment. Patients who received at least one cycle of T-DXd and/or SG are included. Immunohistochemical markers may be determined locally. Treatment with T-DXd and SG is administered per national guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was toxicity rate of each drug | From the initiation of ADC to the date of discontinuation (due to any reason), first documented progression, death from any cause or last contact, throughout study completion, up to 24 months
  Adverse events (AEs) were graded according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0)

SECONDARY OUTCOMES:
progression-free survival (PFS) | From the date of disease progression to the date of death from any cause or last contact, throughout study completion,up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Cooperative Oncology Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No